CLINICAL TRIAL: NCT00978614
Title: Valuation of Dose-Dependent Repeated-Dose Neramexane Effects on Cardiac Repolarisation (QT/QTc Interval Duration) Randomized, Double-Blind, Placebo- and Moxifloxacin-Controlled, Ascending Repeated-Dose, Three-Arm Parallel Design ECG Study in Healthy Adult Subjects
Brief Title: Evaluation of Dose-Dependent Repeated-Dose Neramexane Effects on Cardiac Repolarisation (QT/QTc Interval Duration): Electrocardiogram (ECG) Study in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Priv.-Doz. Dr. med. Georg Golor, Parexel International GmbH
Model: Parallel | Masking: Double
Other Study IDs: MRZ 92579/TI/1006
Record Dates: First submitted 2009-09-10; First posted 2009-09-17 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — neramexane

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (1):
- Neramexane, Placebo, Moxifloxacin (Experimental)
  Interventions: Drug: Neramexane

INTERVENTIONS:
Drug: Neramexane — Dosage form:
  25 mg immediate release [IR] tablets (=15.9 mg neramexane free base)
  37.5 mg IR tablets (=23.9 mg neramexane free base)

SUMMARY:
Primary:

* To assess the effects of ascending repeated-doses of oral [p.o.] neramexane at therapeutic and supra-therapeutic steady-state doses on cardiac repolarisation (QT/QTc interval) in healthy male and female subjects.

Secondary:

* To assess the pharmacokinetics [PK] of neramexane and N-OH neramexane (if a validated method will be available for this metabolite) following repeated daily doses of 50 mg (steady state), 75 mg (steady state) and 87.5 mg (steady state).
* To assess the safety and tolerability of neramexane 50 mg, 62.5 mg, 75 mg and 87.5 mg repeated-dose treatments when gradually up-titrated in healthy subjects.
* To assess the concentration-QT relationship.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subject confirmed on the basis of extensive pre-study screening investigations
* Aged 18 to 45, inclusive
* Body mass index [BMI] of 18-28 kg/m² (inclusive) and a body weight of 50 -<90 kg
* Willing and able to provide written informed consent after having been informed of the requirements and the restrictions of the study
* Female subject of child-bearing potential must agree to use a non-hormonal highly effective method of birth control defined as those which result in a low failure rate when used consistently and correctly, such as sexual abstinence, vasectomized partner, non-hormone releasing intrauterine devices [IUDs].
* A sexually active man, who has not been sterilized surgically, must agree to use together with his female partner a double contraception method during intercourse:

  * IUD or hormonal contraception plus condom or diaphragm or spermicide, or
  * condom plus diaphragm or observe abstinence during the entire clinical study until the Final Examination.

Exclusion Criteria:

* History of clinically relevant allergy or known hypersensitivity to neramexane/memantine/amantadine and their derivatives
* History of clinically relevant allergy or known hypersensitivity to moxifloxacin or any other quinolone antibiotics
* History of clinically relevant allergy or known hypersensitivity to any inactive ingredient in any of the used investigational products or positive control especially quinine
* Any contraindications which are indicated in the current SPC of Avalox®
* Evidence or (family) history of long QT syndrome
* Exposure to another investigational agent within the last two months before Day -1
* Lactating or pregnant female, or female planning to become pregnant during study conduct
* Any evidence of a significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, endocrinological, metabolic (acidosis), psychiatric, neurologic, relevant eye disorder or other diseases at screening
* ECG abnormalities of clinical relevance, in particular abnormal prolongations of QT/QTc-interval (i.e. QTc >450 ms, PQ ≥220 ms)
* Systolic blood pressure <95 mmHg or >140 mmHg or diastolic blood pressure <50 mmHg or >95 mmHg in semi-supine position
* Pulse rate <45 or >100 beats per minute
* History of malignancy
* Any clinically relevant deviation in clinical or laboratory assessment
* Acute or chronic clinically relevant infections
* Current evidence of hypokalemia and/or hypomagnesemia (= below lower limit of laboratory normal range plus 0.3 mmol/L as safety margin)
* History of alcohol or illicit drug abuse
* Alcohol consumption averaging more than 40 g for male and more than 20 g for female subjects daily within the last year
* Alcohol consumption within the last 48 hours prior to Day -1 or illicit drug intake in the 4 weeks prior to Day -1
* Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal products (e.g. cholecystectomy, resections of small or large intestine, febrile conditions, chronic diarrhea, chronic vomiting, endocrine disease severe infections, acute inflammations, etc.)
* Allergy to band aid
* Use of any prescribed drugs in the 4 weeks prior to Day -1
* Regular use of over-the-counter [OTC] drugs (except paracetamol, maximum 1 g/day) in the 4 weeks prior to Day -1
* Occasional use of OTC drugs (except paracetamol, maximum 1 g/day) in the 2 weeks prior to Day -1
* Use of any food, food supplement or medication known to induce or inhibit cytochrome P450 [CYP] 2B6 or any other clinical relevant CYP enzymes within two weeks preceding Day -1 (e.g. grapefruit, St. Johns wort)
* Regular caffeine consumption averaging more than 1 L of coffee and/or tea daily or more than 1 L of caffeine-containing lemonades per day within the last year
* Female subject who employed any form of hormonal contraception within 2 months prior to study Day -1 (e.g. oral contraceptives, hormone releasing IUDs, etc.)
* Consume of xanthine derivates (including coffee, tea, chocolate, etc.) or quinine containing beverages (Bitter Lemon, Tonic Water, etc.) within two days prior to Day -1
* Smoker
* Previous participation in the drug administration phase of this trial
* Blood donation more than 450 mL within 60 days prior to Day -2
* Positive results in any of the serology tests (Human Immunodeficiency Virus [HIV1/2] antibodies, hepatitis B surface antigen, antibodies against hepatitis C virus)
* Positive pregnancy test
* Positive drug screen or alcohol test
* Excessive sports within 3 days before Day -2
* Sauna within 48 hours before Day -2
* Employee or direct relative of an employee of the CRO or Merz Pharmaceuticals
* Evidence or suspicion that the subject might not comply with the study directives and/or that he/she is not reliable or trustworthy
* Evidence or suspicion that the subject is not willing or unable to understand the information that is given to him/her as part of the informed consent, in particular regarding the risks and discomfort to which he/she would agree to be exposed
* Vulnerable subject (e.g. person kept in detention)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To assess the effects of ascending repeated-doses of oral [p.o.] neramexane at therapeutic and supra-therapeutic steady-state doses on cardiac repolarisation (QT/QTc interval) in healthy male and female subjects. | steady state, therapeutic dose

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International GmbH, Berlin, Germany